CLINICAL TRIAL: NCT04098263
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation, Safety and Pharmacokinetic Study of LMN-101 in Healthy Volunteers
Brief Title: Safety and Pharmacokinetic Study of LMN-101 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lumen Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAM01
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Campylobacter Jejuni Infection

STUDY DESIGN:
Intervention Model Description: Part A: Open Label Part B: Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part B: Identical-appearing placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part B: Cohort 1 (Active Comparator): 300 mg PO TID given as a single 300-mg capsule of LMN-101 orally three times daily for 28 days
  Interventions: Biological: LMN-101
- Part B: Cohort 2 (Active Comparator): 1000 mg PO TID given as two 500-mg capsules of LMN-101 orally three times daily for 28 days
  Interventions: Biological: LMN-101
- Part B: Cohort 3 (Active Comparator): 3000 mg PO TID given as six 500-mg capsules of LMN-101 orally three times daily for 28 days
  Interventions: Biological: LMN-101
- Part A (Other): 3000 mg PO single dose given as six 500-mg capsules of LMN-101 orally
  Interventions: Biological: LMN-101

INTERVENTIONS:
Biological: LMN-101 — variable heavy chain-derived binding protein designed to bind and inhibit flagellin filament protein of Campylobacter jejuni, delivered in whole spray-dried, encapsulated spirulina biomass

SUMMARY:
This will be a randomized, double-blind, placebo-controlled, dose-escalation study of 3 dose levels of LMN-101. Healthy volunteers will take LMN-101 or placebo orally either as a single dose or at one of three dose levels three times daily over 28 days. Protocol-specified evaluations and procedures will be performed on Days 1-2 and every one-two weeks during dosing. Study observation will continue until 4 weeks after the last dose of study drug.

DETAILED DESCRIPTION:
Healthy volunteers will be sequentially assigned to the following dosing regimens:

Part A:

A single, open-label dose of 3000 mg orally (2 subjects)

Part B:

Subjects will be randomized within a dose regimen to active or placebo treatment:

* 300 mg PO TID (three times daily) given as a single 300-mg capsule of LMN-101 orally three times daily for 28 days (4 subjects) or identical-appearing placebo capsule (2 subjects).
* 1000 mg PO TID given as two 500-mg capsules of LMN-101 orally three times daily for 28 days (4 subjects) or identical-appearing placebo capsules (2 subjects).
* 3000 mg PO TID given as six 500-mg capsules of LMN-101 orally three times daily for 28 days (4 subjects) or identical-appearing placebo capsules (2 subjects).

The primary endpoint is:

• Safety and tolerability of LMN-101.

The secondary endpoints are:

* Peak serum drug concentration following administration of the initial dose and peak serum drug concentration following a course of treatment (if systemic absorption is observed).
* Area under the serum drug concentration versus time curve (AUC) following administration of the initial dose and following a course of treatment (if systemic absorption is observed).
* Induction of serum anti-drug antibodies (if systemic absorption is observed).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 50 years, inclusive, at time of informed consent
2. Willingness to participate after written informed consent obtained
3. Available for all planned clinical visits for physical examinations, blood draws, stool collections
4. General good health, without significant medical illness or abnormal physical examination findings as determined by the PI.
5. Adequate bone marrow reserve, renal and liver function.

   1. Absolute neutrophil count ≥ 1.5 x 10e9/L
   2. Lymphocyte count < 6.0 x 10e9/L
   3. Platelet count ≥ 150 x 10e9/L
   4. Hemoglobin ≥ 110 g/L
   5. Estimated glomerular filtration rate ≥ 40 mL/min/1.73 meter squared
   6. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 3x upper limit of normal (ULN)
   7. Total bilirubin ≤ 1.5x ULN
   8. Serum albumin ≥ 28 g/L
6. Females of childbearing potential should be using and committed to continue using one of the following acceptable birth control methods:

   1. Sexual abstinence (inactivity) or exclusively same-sex partner for 1 month prior to screening through study completion; or
   2. Intrauterine device (IUD) in place for at least 1 month prior to study through study completion; or
   3. Stable hormonal contraception for at least 1 month prior to study through study completion; or
   4. Surgical sterilization (vasectomy) of male partner at least 6 months prior to study.
7. To be considered of non-childbearing potential, females should be surgically sterilized (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 2 months prior to study) or be post-menopausal and at least 3 years since last menses.
8. Male participants must use condoms during the study and through study completion.

Exclusion Criteria:

1. Treatment with an experimental compound within 30 days.
2. Treatment within 30 days or planned use within the study period with immunomodulator or immunosuppressant agent.
3. Pregnancy or breastfeeding.
4. Presence of any of the following clinical conditions:

   1. History of one or more of the following: cardiac insufficiency (NYHA III/IV), uncontrolled cardiac arrhythmias, unstable ischemic heart disease, or uncontrolled hypertension (systolic blood pressure > 170 mmHg or diastolic blood pressure > 110 mmHg).
   2. History of venous thromboembolic disease within 12 months, myocardial infarction, or cerebrovascular accident.
   3. Unstable pulmonary, renal, hepatic, endocrine or hematologic disease.
   4. Gastrointestinal disorder requiring ongoing care by a physician.
   5. Autoimmune disease, mixed connective tissue disease, scleroderma, polymyositis, or significant systemic involvement secondary to rheumatoid arthritis.
   6. Evidence of active malignant disease, malignancies diagnosed within the previous 5 years, or breast cancer diagnosed within the previous 5 years (except skin cancers other than melanoma).
   7. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other opportunistic infections; or major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks.
   8. Positive serology for human immunodeficiency virus (HIV) infection or history of other immunodeficiency illness.
   9. Positive serology results for hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV)
   10. Significant neuromuscular disease or neuropathy
   11. Psychiatric condition
   12. Alcohol or illicit drug abuse/dependency or positive urine toxicology screen for drugs of abuse other than marijuana. Alcohol and tobacco consumption are permitted.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Griffin, MBBS, Principal Investigator — Nucleus Network
Locations (1):
- Royal Brisbane & Women's Hospital, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo group
Period: Overall Study
Arm/Group | Part A | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3 | Placebo
Started | 2 | 4 | 5 | 4 | 6
Completed | 2 | 4 | 4 | 4 | 6
Not Completed | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo identical appearing capsule orally three times daily for 28 days
- Total: Total of all reporting groups
Arm/Group | Part A | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3 | Placebo | Total
Number analyzed (Participants) | 2 | 4 | 5 | 4 | 6 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 5 | 4 | 6 | 21
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (4.2) | 30.3 (8.5) | 32.4 (11.8) | 41 (2.6) | 36.7 (9.8) | 35.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 2 | 5 | 14
  Male | 1 | 1 | 2 | 2 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5 | 3 | 5 | 18
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 5 | 3 | 5 | 17
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 2 | 4 | 5 | 4 | 6 | 21
Baseline Count of AEs [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Adverse Events
Description: Counts of participants with adverse events
Time Frame: Day 1 to Day 56
Measure: Count of Participants; unit: Participants
Arm/Group | Part A | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3 | Placebo
Number analyzed (Participants) | 2 | 4 | 5 | 4 | 6
Participants | 0 | 1 | 3 | 1 | 3

ADVERSE EVENTS:
Time Frame: 56 days
Groups:
- Placebo: Placebo identical appearing capsules orally three times daily for 28 days
Arm/Group | Part A | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/5 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/5 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 0/2 | 1/4 | 3/5 | 1/4 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=2) | Part B: Cohort 1 (N=4) | Part B: Cohort 2 (N=5) | Part B: Cohort 3 (N=4) | Placebo (N=6)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menstruation Delayed (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT04098263/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT04098263/SAP_001.pdf